CLINICAL TRIAL: NCT03850769
Title: Prospective Phase II Single-arm Study of Neoadjuvant Nab-Paclitaxel and S-1 in Patients With Borderline Resectable Pancreatic Cancer
Brief Title: Neoadjuvant Nab-Paclitaxel and S-1 in Borderline Resectable Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-1752
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Borderline Resectable Pancreatic Cancer
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nab-paclitaxel and S-1 (Experimental): neoadjuvant chemotherapy with Nab-paclitaxel and S-1, repeat every 21 days for 4 cycles.
  Interventions: Drug: nab-paclitaxel and S-1

INTERVENTIONS:
Drug: nab-paclitaxel and S-1 — Nab-Paclitaxel: 120 mg/m2 d1, 8, S-1: Body surface area < 1.25 m2, 80 mg/d; Body surface area ≥ 1.25 m2 < 1.50 m2, 100 mg/d; Body surface area ≥1.5 m2, 120 mg/d; Bid, d1-14;

SUMMARY:
This study was a single-arm multicenter prospective phase II clinical study, designed to evaluate the efficacy and safety of neoadjuvant nab-paclitaxel combined with S-1 in patients with borderline resectable pancreatic cancer. A total of 60 subjects who meet the criteria will receive neoadjuvant chemotherapy of nab-paclitaxel and S-1, for a maximum of 4 cycles prior to pancreatectomy. The primary endpoint is R0 resection rate, the secondary endpoints include overall survival and response rate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have good compliance, can understand the research process of this study, and sign a written informed consent
2. Patients with pathologically confirmed pancreatic adenocarcinoma.
3. Patients who have not received prior chemotherapy, radiotherapy or other systematic treatment for pancreatic cancer;
4. Patients with borderline resectable pancreatic cancer ( NCCN Version 1，2019 criteria).
5. ECOG PS 0-1;
6. Tumor size is measurable according to RECIST1.1 criteria
7. Expected survival over 3 months;
8. Bone marrow function: neutrophils≥1.5x109/L, platelets ≥100x109/L, hemoglobin≥ 90g/L;
9. Liver and kidney function: serum creatinine≤1.5ULT; AST and ALT≤ 2.5 ULT; total bilirubin ≤ 1.5 ULT;
10. No contraindications to the use of S-1 and nab-paclitaxel.

Exclusion Criteria:

1. ≥ Grade 2 existing peripheral neuropathy;
2. Any other malignancy within 5 years prior to enrollment, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, bladder, or nonmelanomatous skin cancer.
3. Active, uncontrolled infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate treatment.
4. Severe, active co-morbidity, defined as follows:

   Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months Transmural myocardial infarction within the 6 months of study registration Uncontrolled hypertension, diabetes or arrhythmia. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization.
5. Not able to take medicine orally.
6. Pregnancy or lactation, and women of childbearing age who refused to take appropriate contraceptive measures during the course of this study;
7. Participation in other clinical trial within 30 days before the first dose of the drug;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 3 years
  proportion of patients who achieved R0 resection

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided